CLINICAL TRIAL: NCT07334431
Title: Fruquintinib Combined With Trastuzumab and XELOX as First-line Treatment in Patients With HER2-positive Advanced Gastric or Gastroesophageal Junction Adenocarcinoma: an Open-label, Single-arm, Single-center Phase Ib/II Clinical Study
Brief Title: Fruquintinib Combined With Trastuzumab and XELOX as First-line Treatment in Patients With HER2-positive Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-134-001
Record Dates: First submitted 2025-04-11; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Gastric Adenocarcinoma; Gastric (Stomach) Cancer; GEJ Adenocarcinoma; HER2-positive Gastric Cancer; First-line Therapy; Fruquintinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib＋trastuzumab + XELOX (Experimental)
  Interventions: Drug: fruquintinib＋trastuzumab + XELOX

INTERVENTIONS:
Drug: fruquintinib＋trastuzumab + XELOX — phase Ib: fruquintinib (3+3 dose escalation design): L1: 2 mg/d, L2: 3 mg/d, L3: 4 mg/d, qd po, D1-14, Q3W; XELOX regimen: Oxaliplatin: 130mg/m2, ivgtt 2h, D1, Q3W; Capecitabine: 1000 mg/m2, bid, D1-D14, Q3W; trastuzumab: 8 mg/kg loading dose and then 6 mg/kg maintenance dose, IV, D1, Q3W; phase II: fruquintinib: RP2D; XELOX regimen: Oxaliplatin: 130mg/m2, ivgtt 2h, D1, Q3W; Capecitabine: 1000 mg/m2, bid, D1-D14, Q3W; trastuzumab: 8 mg/kg loading dose and then 6 mg/kg maintenance dose, IV, D1, Q3W. After 6-8 cycles of combination therapy, trastuzumab plus fruquintinib plus capecitabine was given as maintenance therapy until disease progression, death or intolerable toxicity.

SUMMARY:
This study was designed to evaluate the safety and efficacy of fruquintinib plus trastuzumab, and XELOX as first-line treatment for HER2-positive advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood the study and voluntarily signed the informed consent;
* 18-75 years old (including 18 and 75 years old);
* Pathologically determined advanced gastric or gastroesophageal junction adenocarcinoma;
* No previous anti-tumor treatment for metastatic diseases;
* HER2 positive;
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 3 months;
* At least one measurable lesion according to RECIST version 1.1;
* The functions of vital organs met the following requirements (Blood components and cell growth factors were not allowed within 14 days before enrollment):

  * Absolute neutrophil count ≥1.5×109/L;
  * Platelet ≥100×109 /L;
  * Hemoglobin ≥90g/L;
  * Total bilirubin < 1.5 ULN;
  * ALT and/or AST < 1.5 ULN ;
  * Serum creatinine (Cr) <1.5×ULN;
  * Endogenous creatinine clearance ≥50ml/min;
* Female patients of childbearing age should take effective contraceptive measures;
* Good compliance, cooperate with follow-up.

Exclusion Criteria:

* Failure to comply with the study protocol or study procedure;
* Previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors, chemotherapy or immune checkpoint inhibitors;
* Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
* Known presence of symptomatic central nervous system metastasis or brain metastases;
* Had autoimmune disease or history of autoimmune disease within 4 weeks before enrollment;
* Previously received allogeneic bone marrow transplantation or organ transplantation;
* Uncontrolled malignant ascites (defined as ascites that cannot be controlled by diuretics or puncture as determined by the researcher);
* Severe cardiovascular disease, including unstable angina pectoris or myocardial infarction, occurs within 6 months before the start of study treatment;
* Subjects who are allergic to the investigational drug or any of its adjuncts;
* Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;
* International Standardized Ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN;
* The investigator identified clinically significant electrolyte abnormalities;
* Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
* Poorly controlled diabetes mellitus was present before enrollment (fasting glucose concentration ≥CTCAE level 2 after formal treatment);
* Had any disease or condition prior to enrollment that affected drug absorption, or the patient could not take fruquintinib orally;
* Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unresectosed tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
* Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months >30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks >5 mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure >Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) <50%;
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure >Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) >50%;
* Unmitigated toxicity higher than CTCAE v5.0 grade 1 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;
* Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
* Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 14 days before enrollment;
* Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk；
* Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume > 1.0g;
* Complications require long-term treatment with immunosuppressants or systemic or local use of immunosuppressive corticosteroids (> 10mg/ day prednisone or other therapeutic hormone);
* Investigators believe that the patient has any other conditions that are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 doses (RP2Ds) | When the first cycle of treatment is completed（approximately 21 days）
  To determine the recommended phase 2 dose of fruquintinib, according to the dose limiting toxicities (DLTs).
PFS | Up to 3 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
OS | Up to 3 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
ORR | Up to 3 years
  ORR is defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) per RESISTv1.1.
DCR | Up to 3 years
  DCR is defined as the percentage of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD) per RESISTv1.1.

OTHER OUTCOMES:
Exploratory endpoints | Up to 3 years
  To investigate the correlations between PD-L1, CD-47B, HER2 expression and immune cell infiltration with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Lv, Principal Investigator — Henan Cancer Hospital (Affiliated Cancer Hospital of Zhengzhou University)
Locations (1):
- Henan Cancer Hospital (Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20728210/